CLINICAL TRIAL: NCT03147898
Title: Characterization of Humoral and Cell-Mediated Immune Responses Following a Booster Dose of Pertussis Vaccine
Brief Title: Observational Study Describing the Immune Profile Induced By Pertussis Vaccines
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: NGB00001; U1111 1183 5461 (Other: WHO)
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Whooping Cough; Pertussis
Keywords: Whooping cough; Pertussis
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood draw
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Toddlers: Non-intervention observational study. Toddlers will receive wP-containing combination vaccine as part of the national immunization schedule
- Group 2: Toddlers: Non-intervention observational study. Toddlers will receive an aP-containing combination vaccine as part of the national immunization schedule.
- Group 3: Preschooler: Non-intervention observational study. Preschoolers will receive a wP-containing combination vaccine as part of the national immunization schedule.
- Group 4: Preschooler: Non-intervention observational study. Preschoolers will receive an aP-containing combination vaccine as part of the national immunization schedule.

SUMMARY:
This is an observational study designed to describe the immune profile of toddlers and preschoolers with acellular priming after receiving a booster dose of pertussis vaccine.

ELIGIBILITY:
Inclusion Criteria:

An individual must fulfill all of the following criteria in order to be eligible for study enrollment:

Toddler Cohort:

* Aged 15 to 24 months on the day of (V01)
* Has received 3 doses of a licensed pertussis-containing vaccine for a priming series during infancy in accordance with the recommendations of the NIP or his / her primary care physician
* Has written documentation (e.g., immunization record, physician's certificate, vaccination unit registry) available to verify the receipt of 3 doses of a licensed pertussis-containing infant vaccines as per national immunization schedule
* ICF has been signed and dated by the subject's parent(s) / legally acceptable representative(s) and, if required, an independent witness, in accordance with local regulations
* Planned receipt of routine pertussis booster vaccine, preferably, on same date as, and no more than 2 days following, V01
* Participant and parent / legally acceptable representative are able to attend all scheduled visits and to comply with all study procedures

Preschooler Cohort:

* Aged 48 to 59 months on the date of V01
* Has received 4 doses of pertussis-containing combination vaccines as per national immunization schedule

Exclusion Criteria:

An individual fulfilling any of the following criteria is to be excluded from study enrollment:

* Participation at the time of study enrollment or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the study or planned receipt of any vaccine (other than a booster pertussis vaccine) between V01 and V03a
* Receipt of immunoglobulins, blood, or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months, or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks) within the preceding 3 months
* History of clinically- or laboratory-confirmed pertussis as per the WHO recommended case definition
* Bleeding disorder, verbal report of thrombocytopenia, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating venipuncture, in the opinion of the investigator
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (in the opinion of the investigator) or febrile illness (temperature ≥ 38.0°C) at physical examination on V01 of the study. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Receipt of oral or injected antibiotics therapy within the 72 hours preceding the first blood draw. (Topical antibiotics and antibiotic drops are not included in this exclusion criterion).
* Identified as a natural or adopted child of the Investigator or an employee with direct involvement in the proposed study

Ages: 15 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy subjects aged 15 to 59 months
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
Anti Pertussis antibody concentrations pre and post vaccination | Day 30 post vaccination
  The change in antibody concentrations will be measured from pre to post vaccination
Change in magnitude of T-cell responses to pertussis-containing combination vaccines over time | Day 30 post vaccination
  The change in cell mediated immune responses will be evaluated from pre to post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Officer, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Investigational Site, Mexico City, Mexico
- Investigational Site, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com